CLINICAL TRIAL: NCT06801873
Title: Determining the Fingerprint of Endotoxin Tolerance
Acronym: 100LPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL68166.091.18; 2018-4983 (Other: METC Oost Nederland (Ethical Review Board))
Record Dates: First submitted 2025-01-10; First posted 2025-01-30 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Endotoxemia; Sepsis; Systemic Inflammation; Immunosuppresion
Keywords: Systemic inflammation; Human endotoxemia; Sepsis; Immunosuppression; endotoxin tolerance; Genomics; Transcriptomics
MeSH Terms: conditions — Endotoxemia; Sepsis | interventions — Endotoxins; Lipopolysaccharides

STUDY DESIGN:
Intervention Model Description: This study aims to identify the genomic and transcriptomic factors linked to the development of endotoxin tolerance in vivo. To this end, all subjects will be intravenously challenged with endotoxin (2 ng/kg LPS) to evoke a transient systemic inflammatory response and subsequent development of endotoxin tolerance, which will be quantified by the response upon the second endotoxin challenge one week later. LPS is used as a challenge agent and is a non-invenstigational product, all study participants will receive the challenge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LPS (Experimental): All healthy subjects (male/female) are challenged with endotoxin (LPS) twice.
  Interventions: Other: Endotoxin (E. coli O:113, Reference Endotoxin)

INTERVENTIONS:
Other: Endotoxin (E. coli O:113, Reference Endotoxin) — Intravenous administration of 1 ng/kg (total body weight) endotoxin (Lot no. 94332B1; List Biological Laboratories, Campbell, USA). This is a non-investigational product. Endotoxin is used as challenge agent to achieve a controlled inflammatory state.
  Other Names: LPS; Lipopolysaccharide

SUMMARY:
An explorative, prospective study in 100 healthy volunteers who will be challenged with endotoxin twice to identify SNPs and transcripts that are associated with the degree of endotoxin tolerance

DETAILED DESCRIPTION:
Sepsis remains the number one cause of death in the ICU and incident rates are rising. The focus of sepsis research has shifted away from the hyperinflammatory phase towards the detrimental role of immunosuppression, a phenomenon known as "sepsis-induced immunoparalysis". Because to a high level of heterogeneity and a lack of appropriate biomarkers, a much-warranted precision medicine approach is not possible. The identification of novel biomarkers for sepsis-induced immunoparalysis is also hampered by the extreme heterogeneity of the patient population. Experimental human endotoxemia is a highly standardized, controlled and reproducible model, which results in the development of endotoxin tolerance, an immunologic state capturing many hallmarks of sepsis-induced immunoparalysis. This study aims to identify genomic and transcriptomics biomarkers of endotoxin tolerance. Ultimately, this will lead to the identification of novel biomarkers for the early identification of patients who are prone to develop sepsis-induced immunoparalysis, and facilitate precision medicine for this highly vulnerable group. Primarily, the investigators aim to identify SNPs and transcripts that are associated with the degree of endotoxin tolerance. To increase the chances of success, the genomic and transcriptomic data obtained in vivo will be integrated with data obtained by a previously performed in vitro study. Secondary objectives include SNPs and transcripts associated with the inflammatory response, and epigenomic changes, metabolites, and proteins associated with the inflammatory response and the degree of endotoxin tolerance. Furthermore, the investigators will explore the role of gender and sex hormones in the inflammatory response and endotoxin tolerance, as well as the relationship between ex vivo and in vivo inflammatory responses. This is an explorative, prospective study in 100 healthy volunteers who will be challenged with endotoxin twice. The study takes place at the research unit of the department of Intensive Care Medicine of the Radboud University Medical Center, Nijmegen.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 and ≤35 yrs
* Male
* Healthy (as confirmed by medical history, examination, ECG, blood sampling)

Exclusion Criteria:

* Use of any medication
* Smoking
* History or signs of atopic syndrome (asthma, rhinitis with medication and/or eczema)
* Known anaphylaxis or hypersensitivity to the non-investigational products or their excipients.
* History or signs of hematological disease (bone marrow dysfunction):
* Thrombocytopenia (<150*10^9/ml) or anemia (hemoglobin < 8.0 mmol/L)
* Abnormalities in leukocyte differential counts
* History, signs or symptoms of cardiovascular disease, in particular:
* Previous spontaneous vagal collapse
* History of atrial or ventricular arrhythmia
* Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrioventricular block or a complete left bundle branch block
* Hypertension (defined as RR systolic > 160 or RR diastolic > 90)
* Hypotension (defined as RR systolic < 100 or RR diastolic < 50)
* Renal impairment (defined as plasma creatinine >120 μmol/l)
* Liver enzyme abnormalities (above 2x the upper limit of normal)
* Medical history of any disease associated with immune deficiency
* CRP > 20 mg/L, WBC > 12x109/L or < 4 x109/L, or clinically significant acute illness, including infections, within 3 weeks before labeling day
* Previous (participation in a study with) LPS administration
* Any vaccination within 3 months prior to labeling day
* Participation in a drug trial or donation of blood 3 months prior to labeling day
* Recent hospital admission or surgery with general anesthesia (<3 months to labeling day)
* Use of recreational drugs within 21 days prior to labeling day
* Inability to personally provide written informed consent (e.g. for linguistic or mental reasons) and/or take part in the study.
* Unwillingness to be informed about potential chance findings

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
SNPs | 1 hour before the first LPS administration
  Single-nucleotide polymorphisms (SNPs)
Monocyte transcriptomes | 1 hour before and 4 hours after the first LPS administration
  Genome-wide differential mRNA expression of monocytes obtained before and 4 hours after the first endotoxin challenge
Endotoxin tolerance | From 1 hour before the first LPS challenge until 6 hours after the second LPS challenge
  Difference in plasma cytokine concentration profiles upon the first and second endotoxin challenge (including but not limited to TNFα, IL-6, IL-8, and IL-10 all in pg/mL).

SECONDARY OUTCOMES:
Sex hormones | 1 hour before the first LPS administration
  Blood concentrations of estradiol, estrone and testosterone (in pmol/L) and testosteron (in nmol/L)
Gender | Enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Medicine Deparmtent, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Omics data such as SNP/transcriptional/metabolomics data will be shared.
Supporting Information: SAP, Analytic Code
Access Criteria: RNA-seq data for this study will become available on GEO database.